CLINICAL TRIAL: NCT04805346
Title: Remote Ischemic Conditioning for Protection from Treatment-related Cardiotoxicity in Pediatric, Adolescent, and Young Adult Patients Undergoing Anthracycline Chemotherapy
Brief Title: Remote Ischemic Conditioning in Oncology
Acronym: RICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2020-0708
Record Dates: First submitted 2021-03-17; First posted 2021-03-18 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Participants Undergoing Anthracycline Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Therapeutic Group (Experimental): With the patient sitting upright in bed or a chair, the remote ischemic conditioning intervention will consist of 4 automatic cycles of upper arm blood pressure cuff inflation to 200 mm Hg for 5 minutes to induce transient, noninjurious, limb ischemia, followed by cuff deflation for 5 minutes, for a total of 35 minutes (autoRIC®, Cellaegis Devices, Mississauga, ON, Canada). The remote ischemic preconditioning cycles will be performed by trained research personnel prior to each cycle of chemotherapy (total treatments variable based on chemotherapy protocol).
  Interventions: Device: autoRIC®
- Control Group (No Intervention): A control group will undergo a similar procedure, but the cuff will not be inflated.

INTERVENTIONS:
Device: autoRIC® — With the patient sitting upright in bed or a chair, the remote ischemic conditioning intervention will consist of 4 automatic cycles of upper arm blood pressure cuff inflation to 200 mm Hg for 5 minutes to induce transient, noninjurious, limb ischemia, followed by cuff deflation for 5 minutes, for a total of 35 minutes (autoRIC®, Cellaegis Devices, Mississauga, ON, Canada).17 The remote ischemic preconditioning cycles will be performed by trained research personnel prior to each cycle of chemotherapy (total treatments variable based on chemotherapy protocol
  Arms: Therapeutic Group

SUMMARY:
This is a feasibility study at a single site, Cincinnati Children's Hospital Medical Center. Patients undergoing anthracycline chemotherapy for Hodgkin disease and soft-tissue and bone sarcoma who meet eligibility requirements will be approached to participate in the study. The purpose of the study is to determine if performing remote ischemic conditioning (RIC) is feasible in children and young adults receiving anthracycline chemotherapy. The secondary purpose is to describe differences in markers of myocardial injury and stress in children and young adults that receive RIC prior to anthracycline chemotherapy compared to control subjects that receive sham therapy prior to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric, adolescent, or young adult patients, 11 years of age or above.
2. Able to tolerate upper arm blood pressure inflation.

Exclusion Criteria:

1. Previous diagnosis of cardiomyopathy (dilated, hypertrophic, restrictive, myocarditis) or congenital heart disease other than bicuspid aortic valve.
2. Chronic kidney disease as defined as a pre-transplant GFR <80
3. Central line in both upper extremities.
4. Known peripheral vascular disease or vasculitis.
5. Platelet count less than 30,000.
6. Known clotting disorder or hypercoagulability
7. Non-English-speaking patients.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Adverse Effects | 18-24 months from start of enrollment
  Patients with intra-thoracic disease may also receive consolidative radiation that includes portions of the myocardium within the radiation field and thus further increase their risk of developing therapy-related cardiomyopathy. Thus, the development of cardioprotective strategies during therapy for these malignancies is of primary interest to minimize the potential late adverse effects of anthracyclines among the long term survivors of these conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Ryan, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided